CLINICAL TRIAL: NCT02490631
Title: A Randomized Controlled Trial of 2% Chlorhexidine Gluconate Skin Preparation Cloths for the Prevention of Post op Surgical Site Infections in Spine Patients (Decrease SSI or DeSSI)
Brief Title: 2% Chlorhexidine Gluconate Skin Cloths to Prevent SSI in Spine Surgery Patients
Acronym: DeSSI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Sage Products, Inc. (Industry)
Responsible Party: Principal Investigator, Elizabeth Card, Nursing Research Consultant, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 150310
Record Dates: First submitted 2015-06-16; First posted 2015-07-07 (Estimated); Results first posted 2020-02-25 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-02

CONDITIONS: Surgical Site Infections; Post Operative Complication
Keywords: skin flora
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm (No Intervention): Standard of care pre-operative cleansing with soap and water the night before and morning of surgery
- Intervention Arm (Experimental): 2% chlorhexidine gluconate cloths the night before and morning of surgery
  Interventions: Drug: 2% chlorhexidine gluconate cloths

INTERVENTIONS:
Drug: 2% chlorhexidine gluconate cloths — Cleansing twice pre-operatively jawline to toes with 2% chlorhexidine gluconate cloths
  Other Names: SAGE patient preoperative skin preparation cloths
  Arms: Intervention Arm

SUMMARY:
Surgical site infection (SSI) following spinal surgery is a frequent complication and results in higher morbidity, mortality and healthcare costs. SSI following adult spinal surgery is a frequent complication that has been reported to occur in 0.7-12.0% of patients and result in higher postoperative morbidity, mortality and health care costs. Vanderbilt University Medical Center SSI rate is 7%. Treatment for SSI can be challenging often requiring revision surgery, long-term antibiotics, and prolonged hospitalization. The accurate identification of risk factors is thus important in the development of strategies to prevent these potentially devastating infections. This study proposes a randomized, controlled trial of neuro-spine patients of 2% chlorhexidine gluconate skin preparation cloths for the prevention of post op surgical site infections in spine patients.

Use of CHG cloths the night before and morning of surgery (neckline to toes) will affect (decrease rates) of SSI compared to patients who receive routine standard of care (soap and water pre-op, day of surgery and daily post-operative).

DETAILED DESCRIPTION:
Pre-operatively patients scheduled for neurosurgical spine cases will be evaluated and approached for interest, if consenting process completed, patients will be randomized to one of 2 arms in 1:1 through a block randomization table.

Those enrolled into the study arm will receive the CHG cloths and instructions for use from research personal. Those randomized to the control arm will receive standard of care skin cleansing by nursing staff.

All subjects who have signed consent will have a skin swab culture taken the day of screening and prior to cleansing with Chlorhexidine gluconate wipes close to the intended incision line. The investigators will also obtain skin swab cultures at site of incision preoperatively on the day of surgery, post-op day 4 or time of discharge and at the 30 day follow up.

Both groups will be evaluated daily by study personnel for the development of SSI until post-op day 4 or hospital discharge whichever one comes first. After dressing removal, a daily high definition picture will be taken of the incision line to further document signs of SSI development (pictures will not have any patient identifiable information). Additional evaluations will take place at the 30 day (+/- 7 days) post-op visit. Blinded evaluators utilizing the CDC guideline will grade the incision line for presence of SSI. Measured change in skin flora will be performed by comparing skin swab cultures of intervention group versus standard of care group and individual changes pre and post operatively.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for a neuro-spine procedure and have 2 of the following risk factors:

* Diabetic OR
* BMI>30 OR
* ASA>2 OR
* pre-operatively hospitalized OR
* >60 years old OR
* chronic steroids/immunosuppressive medications OR
* prior history of SSI

Exclusion Criteria:

* Unable to consent
* Non English speaking
* Known allergy to any of the ingredients contained in SAGE chlorhexidine gluconate cloths
* Current infection or history of spine infections
* Patients with tumors or intradural spinal pathology.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Abbey DM, Turner DM, Warson JS, Wirt TC, Scalley RD. Treatment of postoperative wound infections following spinal fusion with instrumentation. J Spinal Disord. 1995 Aug;8(4):278-83. doi: 10.1097/00002517-199508040-00003. PMID 8547767
- [Background] Balderston RA, Blumberg K (1991) Infection in spine surgery. In: Balderston RA, An HS (eds) Complications in spinal surgery. WB Saunders, Philadelphia, pp 157-168
- [Background] Glassman SD, Dimar JR, Puno RM, Johnson JR. Salvage of instrumental lumbar fusions complicated by surgical wound infection. Spine (Phila Pa 1976). 1996 Sep 15;21(18):2163-9. doi: 10.1097/00007632-199609150-00021. PMID 8893444
- [Background] Keller RB, Pappas AM. Infection after spinal fusion using internal fixation instrumentation. Orthop Clin North Am. 1972 Mar;3(1):99-111. No abstract available. PMID 5012590
- [Background] Kostuik JP, Israel J, Hall JE. Scoliosis surgery in adults. Clin Orthop Relat Res. 1973 Jun;(93):225-34. doi: 10.1097/00003086-197306000-00022. No abstract available. PMID 4722945
- [Background] Lonstein J, Winter R, Moe J, Gaines D. Wound infection with Harrington instrumentation and spine fusion for scoliosis. Clin Orthop Relat Res. 1973 Oct;(96):222-33. No abstract available. PMID 4584242
- [Background] Roberts FJ, Walsh A, Wing P, Dvorak M, Schweigel J. The influence of surveillance methods on surgical wound infection rates in a tertiary care spinal surgery service. Spine (Phila Pa 1976). 1998 Feb 1;23(3):366-70. doi: 10.1097/00007632-199802010-00016. PMID 9507627
- [Background] West JL 3rd, Ogilvie JW, Bradford DS. Complications of the variable screw plate pedicle screw fixation. Spine (Phila Pa 1976). 1991 May;16(5):576-9. doi: 10.1097/00007632-199105000-00016. PMID 2053001
- [Background] Olsen MA, Mayfield J, Lauryssen C, Polish LB, Jones M, Vest J, Fraser VJ. Risk factors for surgical site infection in spinal surgery. J Neurosurg. 2003 Mar;98(2 Suppl):149-55. PMID 12650399
- [Background] Calderone RR, Garland DE, Capen DA, Oster H. Cost of medical care for postoperative spinal infections. Orthop Clin North Am. 1996 Jan;27(1):171-82. PMID 8539047
- [Background] Davis H. Increasing rates of cervical and lumbar spine surgery in the United States, 1979-1990. Spine (Phila Pa 1976). 1994 May 15;19(10):1117-23; discussion 1123-4. doi: 10.1097/00007632-199405001-00003. PMID 8059266
- [Background] Patel N, Bagan B, Vadera S, Maltenfort MG, Deutsch H, Vaccaro AR, Harrop J, Sharan A, Ratliff JK. Obesity and spine surgery: relation to perioperative complications. J Neurosurg Spine. 2007 Apr;6(4):291-7. doi: 10.3171/spi.2007.6.4.1. PMID 17436915
- [Background] Rihn JA, Lee JY, Ward WT. Infection after the surgical treatment of adolescent idiopathic scoliosis: evaluation of the diagnosis, treatment, and impact on clinical outcomes. Spine (Phila Pa 1976). 2008 Feb 1;33(3):289-94. doi: 10.1097/BRS.0b013e318162016e. PMID 18303461
- [Background] Pull ter Gunne AF, van Laarhoven CJ, Cohen DB. Incidence of surgical site infection following adult spinal deformity surgery: an analysis of patient risk. Eur Spine J. 2010 Jun;19(6):982-8. doi: 10.1007/s00586-009-1269-1. Epub 2010 Jan 12. PMID 20066445
- [Background] Pull ter Gunne AF, Cohen DB. Incidence, prevalence, and analysis of risk factors for surgical site infection following adult spinal surgery. Spine (Phila Pa 1976). 2009 Jun 1;34(13):1422-8. doi: 10.1097/BRS.0b013e3181a03013. PMID 19478664
- [Background] Eiselt D. Presurgical skin preparation with a novel 2% chlorhexidine gluconate cloth reduces rates of surgical site infection in orthopaedic surgical patients. Orthop Nurs. 2009 May-Jun;28(3):141-5. doi: 10.1097/NOR.0b013e3181a469db. PMID 19494763
- [Background] Karki S, Cheng AC. Impact of non-rinse skin cleansing with chlorhexidine gluconate on prevention of healthcare-associated infections and colonization with multi-resistant organisms: a systematic review. J Hosp Infect. 2012 Oct;82(2):71-84. doi: 10.1016/j.jhin.2012.07.005. Epub 2012 Aug 11. PMID 22889522
- [Background] Climo MW, Yokoe DS, Warren DK, Perl TM, Bolon M, Herwaldt LA, Weinstein RA, Sepkowitz KA, Jernigan JA, Sanogo K, Wong ES. Effect of daily chlorhexidine bathing on hospital-acquired infection. N Engl J Med. 2013 Feb 7;368(6):533-42. doi: 10.1056/NEJMoa1113849. PMID 23388005
- [Background] Milstone AM, Elward A, Song X, Zerr DM, Orscheln R, Speck K, Obeng D, Reich NG, Coffin SE, Perl TM; Pediatric SCRUB Trial Study Group. Daily chlorhexidine bathing to reduce bacteraemia in critically ill children: a multicentre, cluster-randomised, crossover trial. Lancet. 2013 Mar 30;381(9872):1099-106. doi: 10.1016/S0140-6736(12)61687-0. Epub 2013 Jan 28. PMID 23363666

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant signed consent, was randomized to the chlorhexidine arm, but their surgery was cancelled, so they did not start the study. There is no data for this subject.
Groups:
- Standard of Care Pre-operative Cleansing: Standard of care pre-operative cleansing with soap and water the night before and morning of surgery
- 2% Chlorhexidine Gluconate: 2% chlorhexidine gluconate cloths the night before and morning of surgery
  2% chlorhexidine gluconate cloths: Cleansing twice pre-operatively jawline to toes with 2% chlorhexidine gluconate cloths
Period: Overall Study
Arm/Group | Standard of Care Pre-operative Cleansing | 2% Chlorhexidine Gluconate
Started | 79 | 78
Completed | 76 | 75
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Pre-operative Cleansing | 2% Chlorhexidine Gluconate | Total
Number analyzed (Participants) | 76 | 75 | 151
Age, Continuous [Mean (Full Range); unit: years] | 63 [57 to 71.25] | 66 [61 to 72] | 64 [57 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 34 | 74
  Male | 36 | 41 | 77
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 76 | 75 | 151

OUTCOME MEASURES:

1. Primary Outcome: Participants With Surgical Site Infection Development at 30 Days Post-operative
Description: Evaluation daily using the CDC guidelines, daily measurements and deidentified photos
Time Frame: post op day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Pre-operative Cleansing | 2% Chlorhexidine Gluconate
Number analyzed (Participants) | 76 | 75
Participants | 5 | 5
Statistical Analysis 1: Comparison: Standard of Care Pre-operative Cleansing vs 2% Chlorhexidine Gluconate; Test type: Superiority; p = 0.456, Chi-squared

2. Secondary Outcome: Number of Participants With Positive or Abnormal Skin Cultures on Day of Surgery, Day of Discharge, 30 Days Post-op
Description: Skin swabs collected on Day of Surgery, Day of Discharge, 30 days post-op
Time Frame: Day of Surgery, Day of Discharge, 30 days post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Pre-operative Cleansing | 2% Chlorhexidine Gluconate
Number analyzed (Participants) | 76 | 75
Participants
  day of surgery | 41 | 7
  day of discharge | 21 | 9
  30 days post-op | 32 | 25
Statistical Analysis 1: Comparison: Standard of Care Pre-operative Cleansing vs 2% Chlorhexidine Gluconate; Test type: Superiority; p = .019, Chi-squared

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Standard of Care Pre-operative Cleansing | 2% Chlorhexidine Gluconate
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/75
Other Adverse Events (participants affected / at risk) | 0/76 | 0/75

LIMITATIONS AND CAVEATS:
larger sample size needed to examine the relationship between normal skin cultures in the Chlorhexidine arm vs control and development of surgical site infections by day 30.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT02490631/Prot_SAP_000.pdf